CLINICAL TRIAL: NCT03813264
Title: Optimizing Outcomes of Dynamic Psychotherapy by the MATRIX: A Preliminary Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Shlomo Mendlovich, director of the Shalvata Mental Health Center, Shalvata Mental Health Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SHA-0013-18
Record Dates: First submitted 2019-01-03; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Psychotherapy; Mental Health; Monitoring
Keywords: MATRIX; ROM (Routine Outcome Measures); mobile-assisted PROMS; managed care
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The proposed study consists of two complementary processes: the first is the routine collection of clinical data using ROM; The second process is MATRIX-based intervention that is expected to improve the course of treatment.
  The study will take place in the clinic complex located at the Shalvata Mental Health Center campus (Shalva clinic, departmental follow-up clinics, day department), and will include 10 therapists (psychiatrists, psychologists, social workers) and 10 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- preliminary arm (Experimental): pairs of patients and their therapists
  Interventions: Other: Routine outcome measures (ROM)

INTERVENTIONS:
Other: Routine outcome measures (ROM) — The proposed study consists of two complementary processes: the first is the routine collection of clinical data using ROM; The second process is MATRIX-based intervention that is expected to improve the course of treatment.
  Other Names: MATRIX (a tool for analysis of therapeutic hours)

SUMMARY:
Mental disorders require therapeutic effort that contains drug components and psychotherapeutic intervention. The latter requires many resources in light of the skill required. Moreover, such intervention is long, and it takes a long time to assess its effectiveness. The proposed study seeks to implement a management system (ie, a system that monitors and intervenes in ineffective and even harmful treatments) for the purpose of optimizing psychotherapies. The system monitors the improvement in patients' condition in treatment using a mobile phone-based system, and when the treatment is ineffective, it recommends correction strategies. The study will help reduce the ineffective or harmful treatment in dynamic psychotherapy, increasing the quality of care the patient receives. And will lead to the optimal utilization of resources in the mental health system.

DETAILED DESCRIPTION:
The purpose of the proposed study is to examine, on a preliminary basis, the feasibility of a monitoring and intervention system that will enable the identification and even improvement of ineffective (and even harmful) hours of therapy in dynamic psychotherapy.

The study will take place in the clinic complex located at the Shalvata Mental Health Center campus (Shalva clinic, departmental follow-up clinics, day department), and will include 10 therapists (psychiatrists, psychologists, social workers) and 10 patients.The duration of the study will be two months. Once the patient and the therapist have signed an informed consent form, they will be integrated into a cellular-based routine outcome monitoring (ROM) that is developed specifically for the present study. This system, which is completely separate from the clinical systems of the Center, is operated after each session by the therapist. Its activation sends an SMS to the patient and to the therapist, in which a referral to a designated and secure site in which questionnaires are administered in order to measure the patient's condition and the assessment of the therapist and the patient regarding the quality of the therapeutic session. In addition, during the entire study period, the hours of treatment will be recorded in a dedicated manual recording device. This is done routinely in many research institutes in Israel and around the world, with the aim of approving the analysis of inefficient or harmful treatment hours. Treatment hours based on ROM data that have a negative effect (ie, evaluated negatively by the patient) will be transcribed by the therapist, and will undergo full MATRIX analysis. In each treatment pair, an analysis of up to two hours will be possible throughout the four months of the study. This analysis includes the conversion of the text to MATRIX codes, 3-letter codes that mark the section speaker (patient or therapist), the subject of the section (patient, therapist, or both) and its character (whether it deals with the ability to experience [ , Or the relationship between experiences [interrelation]). The coding will be performed by the principal investigator or by the secondary investigator. After the encoding analysis, a MATRIX-based feedback will be given by the Principal Investigator to the therapist, in which the recommendations of the analysis will be submitted.

The proposed study combines routine conventional follow-up practices (ROM) in psychotherapy with innovative analysis tools (MATRIX), and seeks to be a first and significant step in addressing the urgent need to implement managed care in psychotherapy. This has far-reaching implications for the management of mental health care in community, clinic, day care and hospitalization units.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (patients / therapists) over the age of 18.
* had agreed to participate in the study.
* eligible for psychotherapeutic treatment.
* treated with the attending clinician for at least two months.
* treated/treating with dynamic psychotherapeutic treatment only.

Exclusion Criteria:

* Patients who (due to cognitive impairment, language gaps, etc.) are unable to complete a questionnaire with little help.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
implementation of patient/therapist mobile phone based routine monitoring tools in public psychiatric services. | 12 months
  high adherence rate of routine mobile based measures
efficiency of a platform that combine monitor and intervene clinical practice | 12 months
  outcome of psychotherapeutic treatments based on the collection of routine outcomes [ROM] and analysis of MATRIX as measured by the OQ-45 (the most common outcome questionnaire in psychotherapy).

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata Mental Health center, Hod HaSharon, Israel

IPD SHARING:
Plan to Share IPD: No